CLINICAL TRIAL: NCT06434103
Title: An Open, Multicenter Phase I/II Trial of SHR-A1921 in Combination With Adebrelimab and SHR-8068 With or Without Carboplatin in the Treatment of Advanced NSCLC
Brief Title: Clinical Study of SHR-A1921 Combined With Adebrelimab and SHR-8068 With or Without Carboplatin in the Treatment of Advanced NSCLC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1921-205
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Advanced Non-small Cell Lung Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1921 combined with Adebrelimab and SHR-8068 with or without carboplatin (Experimental)
  Interventions: Drug: SHR-A1921；Adebrelimab；SHR-8068；carboplatin

INTERVENTIONS:
Drug: SHR-A1921；Adebrelimab；SHR-8068；carboplatin — SHR-A1921:Specified dose on specified days. SHR-8068: Specified dose on specified days. Adebrelimab: Specified dose on specified days. Carboplatin:Specified dose on specified days.

SUMMARY:
A trial to evaluate the tolerability and efficacy of SHR-A1921 in combination with adbelizumab and SHR-8068 with or without carboplatin in patients with advanced non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to join the clinical study, and sign the informed consent, compliance is good, can cooperate with follow-up;
2. Aged 18-75 at the time of signing the informed consent;
3. Histologically or cytologically confirmed patients with locally advanced or metastatic non-cellular lung cancer who are not eligible for surgical resection or radical concurrent chemoradiotherapy;
4. At least one measurable lesion consistent with RECIST v1.1;
5. ECOG PS score: 0-1;
6. The organ function level is good;

Exclusion Criteria:

1. Untreated (radiation or surgery) central nervous system metastasis, or accompanied by meningeal metastasis, spinal cord compression, etc.;
2. Uncontrolled pleural effusion, pericardial effusion, or peritoneal effusion with clinical symptoms;
3. Previous or co-existing malignant neoplasms;
4. The presence of any active or known autoimmune disease;
5. Have clinical symptoms or diseases of the heart that are not well controlled;
6. People with past or current interstitial pneumonia/interstitial lung disease;
7. Known allergic reactions to any component of SHR-A1921, Adebrelimab, or severe allergic reactions to other monoclonal antibodies;
8. Have previously received topoisomerase I inhibitors (including but not limited to irinotecan, Topotecan), TROP-2ADC, or ADC drugs containing topoisomerase I inhibitors; Previously received anti-PD-1 /PD-L1 antibody or anti-CTLA-4 antibody treatment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
DLT | 21 days after the first dose
ORR based on RECIST v1.1 assessment. | All enrolled subjects were evaluated every 6 or 9 weeks starting with the first dose, up to 2 years

SECONDARY OUTCOMES:
Adverse event | All informed subjects signed informed consent from the beginning to the end of the safety follow-up period， up to 2 years
DCR based on RECIST v1.1 assessment | All enrolled subjects were evaluated every 6 or 9 weeks starting with the first dose, up to 2 years

IPD SHARING:
Plan to Share IPD: Undecided